CLINICAL TRIAL: NCT05424627
Title: Involvement of Myeloid Derived Suppressor Cells in Systemic Lupus Erythematosus
Brief Title: Myeloid Derived Suppressor Cells in Systemic Lupus Erythematosus
Acronym: MDSC-SLE
Status: Not yet recruiting | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Thomas MOULINET, MD, Central Hospital, Nancy, France
Other Study IDs: 2022-A00601-42
Record Dates: First submitted 2022-06-15; First posted 2022-06-21 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Systemic Lupus Erythematosus
Keywords: myeloid derived suppressor cells
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Collection of peripheral blood mononuclear cells for functionnal and flow cytometry analysis.
  Collection of serum for cytokine level assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Systemic Lupus Erythematosus (SLE) is a chronic invalidating chronic condition, with potential articular, cutaneous, renal, and neurologic involvement. Its pathophysiology is complex, and involves genetic, environmental and hormonal factors, leading to tolerance rupture. Among regulatory cells, Myeloid Derived Suppressor Cells (MDSCs) have been described as being increased during SLE, furthermore during flares. MDSCs are defined phenotypically as being HLA-DR-CD3-CD19-CD33+CD11b+, and either CD14+ (Monocytic MDSCs), CD15+ (Granulocytic MDSCs), or CD14-CD15- (Early-stage MDSCs). However, data regarding their immunosuppressive properties are conflicting, some studies identifying regulatory properties, while other have demonstrated a pro-inflammatory involvement through the induction of Th17 lymphocytes.

The objectives of this study is to assess the involvement of MDSC in SLE through accurate phenotypical and functional assessment, as well as characterizing their immunometabolic profile, and to identify innovative therapeutic strategies.

DETAILED DESCRIPTION:
Systemic Lupus Erythematosus (SLE) is a chronic invalidating chronic condition, with potential articular, cutaneous, renal, and neurologic involvement. Its pathophysiology is complex, and involves genetic, environmental and hormonal factors, leading to tolerance rupture. Among regulatory cells, Myeloid Derived Suppressor Cells (MDSCs) have been described as being increased during SLE, furthermore during flares. MDSCs are defined phenotypically as being HLA-DR-CD3-CD19-CD33+CD11b+, and either CD14+ (Monocytic MDSCs), CD15+ (Granulocytic MDSCs), or CD14-CD15- (Early-stage MDSCs). However, data regarding their immunosuppressive properties are conflicting, some studies identifying regulatory properties, while other have demonstrated a pro-inflammatory involvement through the induction of Th17 lymphocytes.

To gain insight into the involvement of MDSC in SLE, both deep phenotypical characterization of MDSC and functional assessment will be performed, as well as immunometabolic characterization. This data will be correlated to the clinical presentation and activity of SLE.

ELIGIBILITY:
Inclusion Criteria:

* Active systemic lupus erythematosus (SLEDAI > or = 1)
* Written informed consent

Exclusion Criteria:

* Chronic or acute infection
* Other active auto-immune condition
* Active cancer
* Age below 18

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with active SLE
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-07-15 (Estimated); Primary Completion 2026-07-15 (Estimated); Study Completion 2027-01-15 (Estimated)

PRIMARY OUTCOMES:
MDSC percentage among total PBMC | Baseline
  Correlation between MDSC percentage among total PBMC and Clinical activity of SLE (SLEDAI score)
MDSC percentage among total PBMC | 3 months
  Correlation between MDSC percentage among total PBMC and Clinical activity of SLE (SLEDAI score)
MDSC percentage among total PBMC | 6 months
  Correlation between MDSC percentage among total PBMC and Clinical activity of SLE (SLEDAI score)
MDSC percentage among total PBMC | Between 9 and 24 months if patient experience relapse during follow-up
  Correlation between MDSC percentage among total PBMC and Clinical activity of SLE (SLEDAI score)

SECONDARY OUTCOMES:
Serum cytokine levels | Baseline
  pro and anti-inflammatory cytokine levels in serum
Serum cytokine levels | 3 months
  pro and anti-inflammatory cytokine levels in serum
Serum cytokine levels | 6 months
  pro and anti-inflammatory cytokine levels in serum
Serum cytokine levels | Between 9 and 24 months if patient experience relapse during follow-up
  pro and anti-inflammatory cytokine levels in serum
MDSC inflammasome activation | Baseline
  flow cytometry assessment of inflammasome activation within MDSCs
MDSC inflammasome activation | 3 months
  flow cytometry assessment of inflammasome activation within MDSCs
MDSC inflammasome activation | 6 months
  flow cytometry assessment of inflammasome activation within MDSCs
MDSC inflammasome activation | Between 9 and 24 months if patient experience relapse during follow-up
  flow cytometry assessment of inflammasome activation within MDSCs
Immunometabolic profile | Baseline
  flow cytometry assessment of metabolic profile of MDSCs
Immunometabolic profile | 3 months
  flow cytometry assessment of metabolic profile of MDSCs
Immunometabolic profile | 6 months
  flow cytometry assessment of metabolic profile of MDSCs
Immunometabolic profile | Between 9 and 24 months if patient experience relapse during follow-up
  flow cytometry assessment of metabolic profile of MDSCs
MDSC subpopulations percentage | Baseline
  flow cytometry assessment of known (Monocytic, Granulocytic, Early-stage) and unknow subpopulations of MDSC
MDSC subpopulations percentage | 3 months
  flow cytometry assessment of known (Monocytic, Granulocytic, Early-stage) and unknow subpopulations of MDSC
MDSC subpopulations percentage | 6 months
  flow cytometry assessment of known (Monocytic, Granulocytic, Early-stage) and unknow subpopulations of MDSC
MDSC subpopulations percentage | Between 9 and 24 months if patient experience relapse during follow-up
  flow cytometry assessment of known (Monocytic, Granulocytic, Early-stage) and unknow subpopulations of MDSC

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Moulinet, Principal Investigator — CHRU de Nancy
Locations (1):
- Thomas Moulinet, Vandœuvre-lès-Nancy, Lorraine, France

IPD SHARING:
Plan to Share IPD: No